CLINICAL TRIAL: NCT03454477
Title: From the Endoscope to the Robot, the Initial Experience of Robotic Thyroidectomy is Summarized
Brief Title: Comparison Between Robotic, Endoscopic and Traditional Open Surgery in Thyroidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Bo Wang,MD, clinical professor, Fujian Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Robotic thyroidectomy
Record Dates: First submitted 2018-02-07; First posted 2018-03-06 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Endoscopy; Robotics; Thyroidectomy; Papillary Thyroid Carcinoma
Keywords: Endoscopy; Robotics; Thyroidectomy; Papillary Thyroid Carcinoma
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- conventional open surgery (Experimental): Patients who met the inclusion criteria were selected for a conventional open surgery procedure for a conventional neck incision for thyroid surgery.
  Interventions: Procedure: conventional open surgery
- endoscopic thyroidectomy (Experimental): Patients who met the inclusion criteria were selected to undergo thyroid surgery via endoscopic thyroidectomy
  Interventions: Procedure: endoscopic thyroidectomy
- robotic thyroidectomy (Experimental): Patients who met the inclusion criteria chose the Da Vinci robot for thyroid surgery.
  Interventions: Device: robotic thyroidectomy

INTERVENTIONS:
Procedure: conventional open surgery — conventional open surgery
  Arms: conventional open surgery
Procedure: endoscopic thyroidectomy — endoscopic thyroidectomy
  Arms: endoscopic thyroidectomy
Device: robotic thyroidectomy — robotic thyroidectomy
  Arms: robotic thyroidectomy

SUMMARY:
Comparison of endoscopic thyroidectomy, robotic thyroidectomy and conventional open surgery, the safety of the operation, the timing of the operation and the complications.

DETAILED DESCRIPTION:
With the further development of endoscopic technique, thyroid surgery of the robot has emerged, which may become a trend of endoscopic technology due to its convenience and accuracy.In this study, the advantages and disadvantages of endoscopic thyroidectomy and robotic thyroid surgery were compared, and the experience in the transition stage of thyroid surgery in robotic and endoscopic thyroidectomy was summarized.

ELIGIBILITY:
Inclusion Criteria:

* Thyroid papillary carcinoma.
* The tumor diameter is less than or equal to 1cm.
* The lymph nodes are limited to the VI level.
* Voluntary choice of endoscopy or robotic surgery.

Exclusion Criteria:

* Patients without beauty needs.
* There is lateral neck or mediastinal lymph node metastasis.
* The tumor invades the nerve and surrounding organs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
operation time | The first day after surgery
  Assess the operation time
recurrent laryngeal nerve palsy | 2 months post operation
  the number of recurrent laryngeal nerve palsy

SECONDARY OUTCOMES:
thyroid volume | The day before the operation
  thyroid volume
cosmetic effect | 2 months post operation
  The satisfaction with cosmetic outcomes was analyzed quantitatively using a scoring system that ranged from 1 to 4(1, extremely; 2, fairly; 3, normal; 4: not at all) that was rated by patients at the outpatient clinic 2 months after the operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Wen-xin ZHAO, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided